CLINICAL TRIAL: NCT03663257
Title: Multicenter Observational Cohort Study to Evaluate Cerebral AneurysmFlow Results in Occlusion
Brief Title: Study to Evaluate Cerebral AneurysmFlow Results in Occlusion
Acronym: CARO
Status: Completed | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: XCY610-130253
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Results first posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Intracranial Aneurysm
Keywords: Interventional Neurology; Aneurysm; Neurology; Radiology; AneurysmFlow
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- AneurysmFlow Observational Cohort: Subjects with unruptured, >5mm saccular aneurysm(s) located in the anterior intracranial circulation and suitable for an endovascular treatment with a Flow Diverter Stent enrolled at the centers participating in this CARO study.
  Interventions: Device: AneurysmFlow

INTERVENTIONS:
Device: AneurysmFlow — AneurysmFlow R1.0 is an approved (CE labeled, cleared in US, Canada and Argentina), software tool intended to provide relevant information on the blood flow in a cerebral aneurysm and its parent artery based on angiography. It provides color coded and vector field representation of a digital subtraction angiography (DSA). It can quantify blood flow rates in the artery based on DSA and 3-D Rotational Angiogram (3DRA) data. It can visualize blood flow patterns in an aneurysm based on DSA data. Specifically, it calculates the Mean Aneurysm Flow Amplitude (MAFA) ratio to measure the volumetric flow rate quotient before and after Flow Diverter Stent (FDS) implantation in the region of interest. It is manufactured by Philips Medical Systems B.V., a Philips Healthcare company.

SUMMARY:
AneurysmFlow R1.0 is an approved (i.e. CE labeled, 510k, Health Canada), software tool intended to provide relevant information on the blood flow in a cerebral aneurysm and its parent artery based on angiography. It calculates the Mean Aneurysm Flow Amplitude (MAFA) ratio to measure the volumetric flow rate quotient before and after Flow Diverter Stent (FDS) implantation in the region of interest.

The current study is a prospective, single arm, observational, multicenter cohort study to assess the prognostic value of the MAFA ratio for predicting full aneurysm occlusion 12 months after flow diverter placement.

DETAILED DESCRIPTION:
AneurysmFlow R1.0 is an approved (CE labeled, cleared in US, Canada and Argentina), software tool intended to provide relevant information on the blood flow in a cerebral aneurysm and its parent artery based on angiography. It provides color coded and vector field representation of a digital subtraction angiography (DSA). It can quantify blood flow rates in the artery based on DSA and 3-D Rotational Angiogram (3DRA) data. It can visualize blood flow patterns in an aneurysm based on DSA data. Specifically, it calculates the Mean Aneurysm Flow Amplitude (MAFA) ratio to measure the volumetric flow rate quotient before and after Flow Diverter Stent (FDS) implantation in the region of interest. It is manufactured by Philips Medical Systems bv., a Philips Healthcare company.

120 subjects with unruptured, >5mm saccular aneurysm(s) located in the anterior intracranial circulation and suitable for an endovascular treatment with a Flow Diverter Stent will be enrolled in the study. The enrollment period is expected to last for 1 year.

Physician investigators participating in this study are expected to follow their normal clinical practice in enrolling, treating and following patients with intracranial aneurysms that are amenable to treatment with flow diverter stents. No additional procedures are required of patients in order to participate in this observational study.

Pre-Screening

Patients presenting with intracranial saccular aneurysm(s) will be evaluated by the neuro interventional team, in accordance with institutional practice, to establish an appropriate treatment plan based on the patient's medical condition and available diagnostic screening procedures prior to recruitment in the study. More than one aneurysm in a single patient may be treated, but only one target aneurysm treated with an FDS device will be considered as part of this study. If treatment of the aneurysm with the FDS is deemed appropriate, the institution's guidelines regarding their ethics committee and informed consent process will be followed.

Screening

After obtaining the consent form(s) approved by the local research ethics board (REB), the principal investigator will screen the potential investigation subjects for the CARO study. The principal investigator or his delegates on the study team will enter data in a pre-designed digital Case Report Form (e-CRF). This will include patient demographics, relevant past medical and surgical history, and specific target aneurysm data along with pre-procedural/screening imaging details.

Only patients who meet all inclusion and none of the exclusion criteria will qualify for this study. The measurement and size of each aneurysm will be verified by the principal investigator. If the size of the aneurysm is acceptable, then it will be included in the study. It is recommended that this measurement should be done within 180 days before the procedure.

Index Procedure and Discharge

The investigator will proceed with standard of care procedures on the day of Index Procedure (i.e. FDS insertion) for the target aneurysm(s). Then, endovascular treatment procedure details should be provided for each eligible patient. Blood flow velocity will be calculated using the dedicated software AneurysmFlow (Philips Healthcare, Best, The Netherlands), which will be installed on standard of care imaging equipment. For this purpose, digital subtraction angiograms will be acquired during the procedure; just before and right after placement of the FDS. Calculation of blood flow velocity will be performed automatically on the AneurysmFlow software. There are no additional devices or medications required for the study. The AneurysmFlow software uses standard-of-care 2D DSA and 3D-RA image sequences to determine this flow information. All raw image sequences will be stored for future reference.

This study will not make any recommendation on patient management or on treatment strategy. Also, this software will not disrupt standard-of-care workflow for the interventionalist.

Follow-Ups (6 and 12 months)

All registry patients treated with FDS are expected to follow their routine post treatment clinical visits, which will include a standard-of-care head imaging (e.g. Computed Tomography Angiography (CTA), Magnetic Resonance Angiography (MRA) and/or DSA) test to classify aneurysm occlusion (i.e. Raymond-Roy Occlusion Classification I) at 6 months (±49 days) and 12 months (±49 days). During the 6 and 12 month follow up visits, patient medical charts will be accessed to collect adverse events (if applicable) and document any post-treatment neurological deterioration (neurological assessment, modified Rankin Scale). De-identified data (i.e. clinical notes, imaging reports etc.) will be entered in the relevant e-CRF sections. All (serious) adverse events (i.e. re-operations, ruptures and deaths) whether or not related to the investigational device will be collected and reported conform local rules and regulations.

The total duration of the study is expected to take approximately 2.5 years. Patient enrollment will take place between September 2018 and September 2019. Each subject will be in the study for 1 year (follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Subject with unruptured, ≥5mm saccular aneurysm(s) located in the anterior intracranial circulation and suitable for an endovascular treatment with a Flow Diverter Stent
* Subject is 18 years of age or older, or of legal age to give informed consent per state or national law.
* Subject is available for clinical follow-ups.

Exclusion Criteria:

* Non-saccular brain aneurysm(s) (i.e. dissecting, fusiform, atherosclerotic, mycotic, bifurcational). Prior aneurysm treatment with either endovascular (stenting, coiling) or surgical (clipping) techniques.
* Endovascular treatment assisted with coils or intracranial stents
* Significant or severe allergy to intra-arterial contrast medium uncontrolled by pre-procedure medications.
* Severe kidney disease (Glomerular Filtration Rate < 60).
* Subjects not willing (or able) to attend post FDS insertion standard-of-care follow up clinic visits requiring DSA, head MRI or CTA imaging.
* Subject participates in a potentially confounding drug or device trial during the course of the study.
* Subject meets an exclusion criteria according to national law (e.g. age, pregnant woman, breast feeding woman).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with age 18 or older, of both genders and all races. Patients are considered to be enrolled in the study after they have signed the informed consent form.
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Hanel, MD, PhD, Principal Investigator — Baptist Medical Center Jacksonville
Locations (4):
- United States (2):
  - Baptist Health, Jacksonville, Florida
  - UMass Medical Center, Worcester, Massachusetts
- ENERI, Buenos Aires, Argentina
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AneurysmFlow Observational Cohort
Started | 132
Completed | 106
Not Completed | 26

BASELINE CHARACTERISTICS:
Population: The Analysis Population is defined as all enrolled subjects that met the eligibility criteria, have the AneurysmFlow measurements recorded pre and post Flow Diverter Stent placement, and have the aneurysm occlusion state (Scale of Roy) available for the 6 month and/or 12 month follow up visit.
Arm/Group | AneurysmFlow Observational Cohort
Number analyzed (Participants) | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.0 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Self-reported Race: American Indian or Alaska Native | 0
  Self-reported Race: Asian | 2
  Self-reported Race: Black or African American | 8
  Self-reported Race: White | 93
  Self-reported Race: Native Hawaiian or Other Pacific Islander | 0
  Self-reported Race: Unknown | 3
Region of Enrollment [Number; unit: participants]
  Canada | 14
  Argentina | 55
  United States | 37
Smoking history [Count of Participants; unit: Participants]
  Never smoked or has not smoked within the last 10 years | 33
  Not a current smoker, but has smoked within the past 10 years | 17
  Current smoker, less than one pack per day | 11
  Current smoker, greater than or equal to one pack per day | 3
  Unknown | 42
Medical history [Number; unit: participants]
  Hyperlipidemia | 18
  Hypertension | 44
  Migraines | 22
Type of presentation [Count of Participants; unit: Participants]
  Incidental | 80
  Symptomatic | 26
Aneurysm measurements [Mean (Standard Deviation); unit: mm]
  Aneurysm maximum height | 6.3 (4.3)
  Aneurysm neck diameter | 4.6 (2.2)
Aneurysm location in Internal Carotid Artery segment [Count of Participants; unit: Participants]
  C1 (Cervical Segment) | 1
  C2 (Petrous Segment) | 1
  C3 (Lacerum Segment) | 0
  C4 (Cavernous Segment) | 16
  C5 (Clinoid Segment) | 14
  C6 (Ophthalmic Segment) | 52
  C7 (Communicating Segment) | 19
  Unknown | 3

OUTCOME MEASURES:

1. Primary Outcome: Prognostic Value of the MAFA (Mean Aneurysm Flow Amplitude) Ratio With Respect to Full Aneurysm Occlusion Within 12 Months
Description: To assess the prognostic value (i.e. c-statistic including confidence intervals) of the MAFA ratio with respect to full aneurysm occlusion (i.e. using the Raymond-Roy Occlusion Classification I on standard-of-care head imaging) 12 months after Flow Diverter Stent placement.
  The objective was evaluated using logistic regression analysis to evaluate the univariate predictive association between the index test (i.e., the MAFA ratio) and complete aneurysm occlusion (i.e., complete occlusion yes/no) at 12 months. The primary endpoint was presented using a Receiver Operating Characteristic (ROC) curve including the c-statistic (also known as the Area Under the Curve (AUC) of the ROC curve) and confidence intervals.
Time Frame: 12 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | AneurysmFlow Observational Cohort
Number analyzed (Participants) | 106
probability | 0.540 [0.400 to 0.680]

2. Secondary Outcome: Prognostic Value of the MAFA Ratio With Respect to Full Aneurysm Occlusion Within 6 Months
Description: To assess the prognostic value (i.e. c-statistic including confidence intervals) of the MAFA ratio with respect to full aneurysm occlusion (i.e. using the Raymond-Roy Occlusion Classification I on standard-of-care head imaging) 6 months after Flow Diverter Stent placement.
  The objective was evaluated using logistic regression analysis to evaluate the univariate predictive association between the index test (i.e., the MAFA ratio) and complete aneurysm occlusion (i.e., complete occlusion yes/no) at 12 months. The endpoint was presented using a Receiver Operating Characteristic (ROC) curve including the c-statistic (also known as the Area Under the Curve (AUC) of the ROC curve) and confidence intervals.
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: probability
Arm/Group | AneurysmFlow Observational Cohort
Number analyzed (Participants) | 106
probability | 0.568 [0.450 to 0.680]

3. Secondary Outcome: Optimal MAFA Threshold
Description: To determine the optimal threshold for the MAFA ratio (to predict full aneurysm occlusion within 12 months), ROC analysis will be performed in combination with net-benefit analysis. Net benefit incorporates estimates of prevalence and misclassification costs, and it is clinically interpretable since it reflects changes in correct and incorrect diagnoses when a new diagnostic test is introduced. The optimal MAFA ratio threshold for clinical decision making is defined as the MAFA ratio where the net benefit is maximized.
  MAFA (Mean Aneurysm Flow Amplitude) = (mean aneurysm flow post / mean aneurysm flow pre) * (mean arterial flow pre / mean arterial flow post)
Time Frame: 12 months
Population: The Analysis Population is defined as all enrolled subjects that met the eligibility criteria, have the AneurysmFlow measurements recorded pre and post Flow Diverter Stent (FDS) placement, and have the aneurysm occlusion state (Scale of Roy) available for the 6 month and/or 12 month follow up visit.
Measure: Number; unit: MAFA ratio
Arm/Group | AneurysmFlow Observational Cohort
Number analyzed (Participants) | 106
MAFA ratio | NA — Based on ROC analysis the net benefit curve does not show a maximum for any MAFA ratio and therefore the optimal MAFA ratio threshold for clinical decision making cannot be determined. This is due to an insufficient number of participants with non-occluded aneurysms, along with the fact that the data from occluded and non-occluded cases were too similar to establish the threshold.

4. Secondary Outcome: Serious Adverse Events
Description: To register serious adverse events (i.e. re-operations, ruptures and deaths).
Time Frame: 12 months
Measure: Number; unit: serious adverse events
Arm/Group | AneurysmFlow Observational Cohort
Number analyzed (Participants) | 132
serious adverse events | 6

ADVERSE EVENTS:
Time Frame: 12 months follow up
Arm/Group | AneurysmFlow Observational Cohort
All-Cause Mortality (participants affected / at risk) | 1/132
Serious Adverse Events (participants affected / at risk) | 4/132
Other Adverse Events (participants affected / at risk) | 4/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AneurysmFlow Observational Cohort (N=132)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Device occlusion (Product Issues) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AneurysmFlow Observational Cohort (N=132)
Chest pain (Cardiac disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Stent stenosis (General disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-06): https://cdn.clinicaltrials.gov/large-docs/57/NCT03663257/Prot_SAP_000.pdf